CLINICAL TRIAL: NCT04681092
Title: Anti-COVID19 AKS-452 Phase I/II VaccinaTion Study
Brief Title: Anti-COVID19 AKS-452 Fusion Protein Vaccine - ACT Study
Acronym: ACT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Akston Biosciences Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL2020-005997-82
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Covid19
Keywords: vaccine; safety; immunogenicity; dose-finding; exploratory efficacy
MeSH Terms: conditions — COVID-19 | interventions — AKS-452 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, combinatorial safety, tolerability and exploratory efficacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- AKS-452 s.c.(A) (Experimental): Subcutaneous injection of pre-defined dose (22,5 ug, 125 uL) single-dose
  Interventions: Biological: AKS-452
- AKS-452 s.c. (B) (Experimental): Subcutaneous injection of pre-defined dose (22,5 ug, 125 uL), two-dose
  Interventions: Biological: AKS-452
- AKS-452 s.c. (C) (Experimental): Subcutaneous injection of pre-defined dose (45 ug, 205 uL), single-dose
  Interventions: Biological: AKS-452
- AKS-452 s.c. (D) (Experimental): Subcutaneous injection of pre-defined dose (45 ug, 250 uL), two-dose
  Interventions: Biological: AKS-452
- AKS-452 s.c. (E) (Experimental): Subcutaneous injection of pre-defined dose (90 ug, 500 uL), single-dose
  Interventions: Biological: AKS-452
- AKS-452 s.c. (F) (Experimental): Subcutaneous injection of pre-defined dose (90 ug, 500 uL), two-dose
  Interventions: Biological: AKS-452
- Phase 2, single-dose injection (Experimental): Subcutaneous injection of selected dose based on phase 1 data, dose (90 ug, 500 uL)
  Interventions: Biological: AKS-452
- Phase 2, two-dose injection (Experimental): Subcutaneous injection of selected dose based on phase 1 data, dose (45 ug, 500 uL) twice.
  Interventions: Biological: AKS-452

INTERVENTIONS:
Biological: AKS-452 — s.c. or i.m. vaccination

SUMMARY:
Combinatorial phase I/II safety, tolerability and immunogenicity single center open-label clinical study of AKS-452 COVID-19 vaccination study

DETAILED DESCRIPTION:
The study is designed as a combinatorial single-center open-label phase I and II clinical study design:

I. a phase I dose-finding and safety / tolerability study combined with, II. a phase II safety / efficacy study on the biological activity of AKS-452 against COVID-19.

To warrant more extensive development towards a phase III clinical study. The study will have a duration of approximately 4 months and will be executed at the University Medical Center Groningen, The Netherlands supported by the subsidizing party Akston Biosciences.

ELIGIBILITY:
Inclusion Criteria:

SARS-CoV-2 serology by Akston (a quantitative anti-SARS-Cov-2 SP/RBD-specific IgG ELISA):

* Undetectable or < 5 μg/mL titer and no known prior SARS-Cov-2 infection

  * Body mass index (BMI) between 19.0 and 30.0 kg/m2, inclusive
  * General good health, without significant medical illness, as determined via physical exam findings, ECG or vital signs
* Note: one retest of vital functions and ECG is allowed within the screening window

  - No clinically significant laboratory abnormalities as determined by the investigator
* Note: one retest of lab tests is allowed within the screening window

  * Informed Consent Form signed voluntarily before any study-related procedure is performed, indicating that the subject understands the purpose and procedures required for the study and is willing to participate in the study
  * Willing to adhere to the prohibitions and restrictions specified in this protocol
  * Non-smoker (including prior smokers having stopped smoking for more than 3 months at time of screening) or non-habitual smoker (habitual smokers are persons who smoke more than 4 cigarettes or other tobacco products on a weekly basis) and agree to not use tobacco products during confinement.
  * Negative alcohol breath test and urine drug screen at screening and upon check-in at the clinical site.
  * Negative hepatitis panel (including hepatitis B surface Ag and anti-hepatitis C virus Abs) and negative human immunodeficiency virus Ab and Ag screens at screening
  * Female subjects should fulfil one of the following criteria:
* At least 1 year post-menopausal (amenorrhea >12 months and/or follicle stimulating hormone >30 mIU/mL) at screening;
* Surgically sterile (bilateral oophorectomy, hysterectomy, or tubal ligation);
* Will use adequate forms of contraceptives from screening to discharge.

  - Female subjects of childbearing potential and male subjects who are sexually active with a female partner of childbearing potential must agree to the use of an effective method of birth control from screening to discharge
* Note: medically acceptable methods of contraception that may be used by the subject and/or partner include combined oral contraceptive, contraceptive vaginal ring, contraceptive injection, intrauterine device, etonogestrel implant, double barrier, sterilization and vasectomy

  - Female subject has a negative pregnancy test at screening and upon check-in at the clinical site.
* Note: pregnancy testing will consist of a serum pregnancy test at screening and urine pregnancy tests at other (dosing) visits, in all women.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Pregnant of breastfeeding females
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, hematologic, rheumatologic, endocrine, autoimmune, or renal disease
* Any laboratory test which is abnormal, and which is deemed by the Investigator(s) to be clinically significant
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol
* Current alcohol/illicit drug/nicotine abuse or addiction: history or evidence of current drug use or addiction (positive drug screen for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, or opiates) or excessive use of alcohol at screening and Day -2.
* Presence of any febrile illness (T > = 38.0°C or lab confirmed viral disease (PCR)) or symptoms suggestive of a viral respiratory infection within 1 weeks prior to vaccination
* Use of corticosteroids (excluding topical preparations for cutaneous or nasal use) or use of immunosuppressive drugs within 30 days before inoculation
* A history of anaphylaxis, history of allergic reaction to vaccine, known allergy to one of the components in AKS-452. Mild allergies without angio-oedema or treatment need can be included if deemed not to be of clinical significance (including but not limited to allergy to animals or mild seasonal hay fever)
* A history of asthma within the past 10 years, or a current diagnosis of asthma or reactive airway disease associated with exercise
* Receipt of a licensed vaccine within 4 weeks prior to viral inoculation
* Received any experimental SARA-CoV-2 vaccine or drug
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to vaccination.
* Receipt of another investigational agent within 30 days or 5 times the product half-life (whichever is longest) prior to vaccination
* Shares household with /works with immunocompromised individual(s), adults with significant cardiopulmonary disease, persons with significant asthma, institutionalized elderly or elderly with functional disability
* Deprived of freedom by an administrative or court order or in an emergency setting - Any condition that in the opinion of the principal investigator (PI) would jeopardize the safety or rights of a person participating in the trial or would render the person unable to comply with the protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Safety / Tolerability | 35 days
  CTCAE-scoring

SECONDARY OUTCOMES:
Immunogenicity | 180 days
  Antibody response COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Schelto Kruijff, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feitsma EA, Janssen YF, Boersma HH, van Sleen Y, van Baarle D, Alleva DG, Lancaster TM, Sathiyaseelan T, Murikipudi S, Delpero AR, Scully MM, Ragupathy R, Kotha S, Haworth JR, Shah NJ, Rao V, Nagre S, Ronca SE, Green FM, Aminetzah A, Sollie F, Kruijff S, Brom M, van Dam GM, Zion TC. A randomized phase I/II safety and immunogenicity study of the Montanide-adjuvanted SARS-CoV-2 spike protein-RBD-Fc vaccine, AKS-452. Vaccine. 2023 Mar 24;41(13):2184-2197. doi: 10.1016/j.vaccine.2023.02.057. Epub 2023 Feb 23. PMID 36842886
- [Derived] Janssen YF, Feitsma EA, Boersma HH, Alleva DG, Lancaster TM, Sathiyaseelan T, Murikipudi S, Delpero AR, Scully MM, Ragupathy R, Kotha S, Haworth JR, Shah NJ, Rao V, Nagre S, Ronca SE, Green FM, Aminetzah A, Sollie F, Kruijff S, Brom M, van Dam GM, Zion TC. Phase I interim results of a phase I/II study of the IgG-Fc fusion COVID-19 subunit vaccine, AKS-452. Vaccine. 2022 Feb 23;40(9):1253-1260. doi: 10.1016/j.vaccine.2022.01.043. Epub 2022 Jan 31. PMID 35115195
- See also: Scientific manuscript phase I clinical study AKS-452 — https://doi.org/10.1016/j.vaccine.2022.01.043